CLINICAL TRIAL: NCT03534687
Title: Role of Exercise in the Prevention and Treatment of RAGE-Mediated Inflammation (RECEPTOR) Trial
Brief Title: Exercise and the Receptor for Advanced Glycation End Products (RAGE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jacob Haus, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00146001; 5R01DK109948-02 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: RAGE; ADAM10; Exercise; sRAGE
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Alzheimer Disease 10; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): Aerobic Exercise (AE) subjects will come in for supervised, aerobic exercise training sessions 5 days a week for 12 weeks. Training will progress from 55% VO2max for week 1 (40 min session), to 60-65% VO2max for week 2 (50 min session), to ~70% VO2max for all other weeks (50 min session). Subjects will perform a warm-up and cool down (~5 min each) that includes stretching exercises. Subjects will wear heart rate monitors during each training session to provide feedback of target heart rate. Intensity, duration, resting and exercise heart rates, and blood pressures will be recorded for each session. Follow-up VO2max tests will be performed at weeks 4 and 8 to monitor progress and adjust AE training intensity.
  Interventions: Behavioral: Aerobic Exercise
- Control Group (No Intervention): During the 12 week control period, subjects are to maintain their normal, daily-living activities. Control group participants will be given the option to enroll in the AE training group after completion of the original Control group trial period.

INTERVENTIONS:
Behavioral: Aerobic Exercise — 12-week supervised aerobic exercise
  Arms: Aerobic Exercise Group

SUMMARY:
This study examines the effects of 12-weeks of aerobic exercise training on the mechanisms driving RAGE-mediated inflammation in type 2 diabetic humans.

DETAILED DESCRIPTION:
Activation of RAGE (receptor of advanced glycation endproducts (AGEs)), via binding of AGEs and other ligands, modulates the development and progression of diabetic complications through persistent and cyclic activation of nuclear factor-kappa beta. Targeting RAGE directly as a therapeutic strategy has largely been unsuccessful. However, RAGE signaling can be interrupted, in vivo, by ADAM10 (a disintegrin and metalloproteinase 10) directed proteolytic cleavage of the RAGE ectodomain, and thus creating a soluble isoform of RAGE (sRAGE) that is released from the cell and appears into the circulation. Maintaining high levels of circulating sRAGE is advantageous as sRAGE will sequester RAGE ligands and prevent RAGE cell signaling.

Although the exact mechanisms of ADAM10 mediated RAGE release remain undefined, calcium related and other signaling (SIRT1) impact ADAM10. Aerobic exercise presents a unique model for mechanistic study of RAGE release as muscle contraction induces robust calcium signaling, activates SIRT1, and provides stimuli for tissue remodeling and resolution of the metabolic profile that drives inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 y
* Type 2 diabetes
* Overweight or obese (BMI 26-44 kg/m2)
* Fluency in English (written and verbal)

Exclusion Criteria:

* Age <40 or >75 y
* BMI <26 or >44 kg/m2
* Existing cardiovascular, cerebrovascular, renal, or hematological disease, or cancer
* Current use of tobacco
* Pregnant or lactating
* Medications that may interfere with study outcomes

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Haus, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise Group | Control Group
Started | 20 | 13
Completed | 13 | 11
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Group | Control Group | Total
Number analyzed (Participants) | 20 | 13 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 7 | 23
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9) | 60 (9) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 13 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 12 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 13 | 33
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.6 (6.0) | 32.6 (5.7) | 33.8 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Quantify the Percentage Change in Basal Circulating sRAGE After 12-weeks of Supervised Aerobic Exercise Training.
Description: Serum will be separated from blood samples collected in vacutainer tubes via centrifugation before and after 12-weeks of aerobic exercise training. sRAGE will be quantified in these serum samples via ELISA (Quantikine, Human RAGE Immunoassay) per manufacture's protocol.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change in sRAGE
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 13 | 13
Percent Change in sRAGE | 24.5 (30.7) | 0.5 (27.2)

2. Secondary Outcome: Quantify the Percentage Change in Basal Muscle RAGE Expression After 12-weeks of Supervised Aerobic Exercise Training.
Description: Basal biopsy derived skeletal muscle RAGE expression will be determined from the vastus lateralis before and after 12-weeks of aerobic exercise training. RAGE expression will be quantified via Western Blot. Muscle samples (~10 mg) will be homogenized and protein concentration will be determined via BCA assay (Pierce). Samples (20 μg protein) will be diluted in SDS buffer, heated at 85 °C for 5 min, resolved via SDS-PAGE (Bio-Rad Laboratories, Hercules, CA) and transferred to a nitrocellulose or PVDF membrane. Blocking will occur for 1 h and primary antibody (RAGE; Abcam, Cambridge, MA) incubation will occur overnight at 4 °C and quantified vs a standard or total protein.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change in basal muscle RAGE
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 11 | 8
percent change in basal muscle RAGE | -14.5 (35.6) | 4.45 (36.8)

3. Secondary Outcome: Quantify the Percentage Change in Aerobic Capacity (VO2max) After 12-weeks of Supervised Aerobic Exercise Training.
Description: Maximal oxygen consumption (VO2max) will be established via indirect calorimetry during an incremental treadmill test (Modified Bruce protocol) before and after 12-weeks of aerobic exercise training. Criteria, such as, rating of perceived exertion >18, respiratory exchange ratio >1.10, no further increase in VO2 despite increasing workloads, heart rate greater than age-predicted maximum, or volitional fatigue will be used to indicate a successful VO2max was achieved.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change in aerobic capacity
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 14 | 12
percentage change in aerobic capacity | 6.9 (6.7) | 0.6 (9.0)

4. Secondary Outcome: Quantify the Percentage Change in Insulin Sensitivity After 12-weeks of Supervised Aerobic Exercise Training.
Description: Insulin sensitivity will be established via calculation of Matsuda Index from glucose and insulin values obtained every 30 minutes during a 75 g Oral GlucoseTolerance Test. Data are represented as percent change. Any change greater than a value of zero indicates an improvement in insulin sensitivity.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change in insulin sensitivity
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 12 | 12
percentage change in insulin sensitivity | 79 (186) | 9 (63)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 12-weeks per participant
Description: clinicaltrials.gov definition
Arm/Group | Aerobic Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 0/20 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03534687/Prot_SAP_000.pdf